CLINICAL TRIAL: NCT06881810
Title: Enhancing Social Skills in Schizophrenia Spectrum Disorders - Two-arm, Double-blind, Randomized Clinical Trial Investigating Oxytocin vs. Placebo as an add-on to an Individualized Psychosocial Treatment (OXY-APS)
Brief Title: Enhancing Social Skills in Schizophrenia Spectrum Disorders - Oxytocin as add-on to Psychosocial Treatment
Acronym: OXY-APS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OXY-APS; 2023-509433-40-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-10; First posted 2025-03-18 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia Spectrum Disorders (SSD)

STUDY DESIGN:
Intervention Model Description: two-arm, double-blind, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Experimental): A single dose of 80 I.U. oxytocin in aerosol form (Syntocinon® nasal spray) is administered via 20 puffs 2 times per week intranasally. 1 ml of Syntocinon nasal spray contains 40 I.U. of oxytocin, with one puff equivalent to 0.1 ml of nasal spray (4 I.U. per spray). To reach the dose of 80 I.U. a total of ten spray puffs per nostril are required (1 ml per Nostril, 2 ml in total). The nasal spray is applied in a sitting position:
  * dose: 80 I.U. = 2 ml Syntocinon® nasal spray (cumulative total dose) is administered as intranasal spray twice a week, 45-75 min. before psychosocial intervention twice a week
  * duration of treatment: 12 weeks
  Interventions: Drug: Oxytocin nasal spray
- Placebo (Placebo Comparator): * 2ml placebo dose is administered twice a week, 45-75 min. before psychosocial intervention twice a week
  * duration of treatment: 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oxytocin nasal spray — Syntocinon® nasal spray is applied according to description in arms section
  Arms: Oxytocin
Other: Placebo — Placebo nasal spray is applied according to description in arms section
  Arms: Placebo

SUMMARY:
Research on schizophrenia spectrum disorders (SSD) patients with social impairment is essential for improving treatment, enhancing the lives of affected individuals, reducing stigma, and advancing our understanding of this complex psychiatric disorder. A clinical trial focusing on the improvement of social skills in SSD has the potential to transform clinical practice and support systems to better meet the needs of those living with SSD. Because of the role of oxytocin in regulating social behaviors and emotions, the investigator hypothesizes that it is beneficial in addressing the social cognition deficits observed in SSD when combined with psychosocial interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 64 years
2. Written informed consent (must be available before enrolment in the clinical trial)
3. ICD-11 diagnosis of schizophrenia or other primary psychotic disorders (6A20-6A25) confirmed by the MINI-DIPS-OA Interview
4. At least one symptom of moderate severity or worse in the PANSS negative subscale (a score ≥ 4 for one or more symptoms from N1-N7 at baseline).
5. In- or outpatient psychosocial treatment on a regular basis at least twice a week during the study
6. Male participants and female participants who are not capable of bearing children or female patients of childbearing potential who use a highly effective birth control method that is medically approved by the health authority at screening.

1. Age 18 to 64 years 2. Written informed consent (must be available before enrolment in the clinical trial) 3. ICD-11 diagnosis of schizophrenia or other primary psychotic disorders (6A20-6A25) confirmed by the MINI-DIPS-OA Interview 4. At least one symptom of moderate severity or worse in the PANSS negative subscale (a score ≥ 4 for one or more symptoms from N1-N7 at baseline). 5. In- or outpatient psychosocial treatment on a regular basis at least twice a week during the study 6. Male participants and female participants who are not capable of bearing children or female patients of childbearing potential who use a highly effective birth control method that is medically approved by the health authority at screening.

Exclusion Criteria:

1. Patients who are not suitable for the study in the opinion of the investigator (including acutely suicidal patients)
2. Coercive treatment at the time of study inclusion
3. Diagnosis of primary substance dependency other than nicotine: exclusion alcohol dependency via AUDIT-screening (Bohn, Babor et al. 1995; Babor et al. 2001) and ICD- 11 criteria (MINI-DIPS-OA); exclusion of other drug dependencies other than alcohol and nicotine: drug screening of urine and ICD-11 criteria (MINI-interview: patient fulfilling early (> 3 months) or sustained (>12 months) remission criteria and/or with low severity of substance use disorder according to MINI (ICD-11) are eligible for the study).
4. Documented intolerance to the study drug or any of its ingredients.
5. Pregnancy (incl. positive urine or blood pregnancy test) / breastfeeding (female patients) or lactating individuals
6. Severe endocrinological disorder besides diabetes
7. Endometriosis
8. Concurrent participation

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Personal and Social Performance Scale (PSP) | from Visit 1 to Visit 4 i.e. 12 weeks
  The main purpose of this clinical trial is to evaluate the efficacy and safety of OXT combined with psychosocial interventions for improving social skills and psychopathology in SSD. We hypothesize a greater absolute PSP score improvement when OXT is administered together with the psychosocial intervention.

SECONDARY OUTCOMES:
Positive and Negative Symptom Scale (PANSS) reduction | from Visit 1 to Visit 4 i.e. 12 weeks
  Due to the expected enhanced social functioning in the OXT group we hypothesize a larger PANSS total score reduction comparing V1 and V4 in the exploratory arm and a linear decrease of total PANSS score over the sequential study visits in both treatment arms, but more pronounced in the exploratory arm.
Clinical Global Impression-Schizophrenia scale (CGI-SCH) reduction | from Visit 1 to Visit 4 i.e. 12 weeks
  Due to the expected enhanced social functioning in the OXT group we hypothesize a larger CGI-SCH reduction comparing V1 and V4 in the exploratory arm and a linear decrease of total CGI-SCH score over the sequential study visits in both treatment arms, but more pronounced in the exploratory arm.
Global Assessment of Functioning (GAF) increase | from Visit 1 to Visit 4 i.e. 12 weeks
  Due to the expected enhanced social functioning in the OXT group we hypothesize a larger GAF increase comparing V1 and V4 in the exploratory arm and a linear increase of GAF total score over the sequential study visits in both treatment arms, but more pronounced in the exploratory arm.
Brief Psychiatric Rating Scale (BPRS) reduction | from Visit 1 to Visit 4 i.e. 12 weeks
  Due to the expected enhanced social functioning in the OXT group we hypothesize a larger BPRS reduction in the exploratory arm and a linear decrease of total BPRS score over the sequential study visits in both treatment arms, but more pronounced in the exploratory arm.
WHO Disability Assessment Schedule (WHODAS 2.0) increase | from Visit 1 to Visit 4 i.e. 12 weeks
  Due to the expected enhanced social functioning in the OXT group we hypothesize a larger increase in WHODAS 2.0 in the exploratory arm.
Personal and Social Performance Scale (PSP) | from Visit 1 to Visit 4 i.e. 12 weeks
  Due to the expected enhanced social functioning in the OXT group we hypothesize a linear increase of total PSP score over the sequential study visits in both treatment arms, but more pronounced in the exploratory arm.
B-CATS improvement | from Visit 1 to Visit 4 i.e. 12 weeks
  We hypothesize a larger improvement across the cognitive domains in the relevant psychometric tests (B-CATS) in the exploratory over the course of the study.
Drop Out Rate | from Visit 1 to Visit 4 i.e. 12 weeks
  We hypothesize a smaller likelihood of discontinuation in the OXT group.

CONTACTS AND LOCATIONS:
Overall Officials: Dusan Hirjak, Prof. Dr., Principal Investigator — Central Institute of Mental Health
Locations (1):
- Central Institute of Mental Health, Department of Psychiatry,, Mannheim, Baden-Wurttemberg, Germany